CLINICAL TRIAL: NCT06056427
Title: An Intermediate Size Patient Population Expanded Access Protocol to Evaluate the Safety and Efficacy of Autologous HB-adMSCs for the Treatment of Patients With Parkinson's Disease
Brief Title: Intermediate Size Expanded Access Protocol Using Autologous HB-adMSCs for the Treatment of Parkinson's Disease
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBPD06
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: HB- adMSCs (Hope Biosciences adipose derived mesenchymal stem cells) — Participants will receive autologous HB-adMSCs through intravenous infusion only, with a treatment duration of 18 weeks, infusion rate 4-5mL/min and total volume of 250 mL Sodium chloride 0.9%. Each participant will receive a total of 6 doses of HB-adMSCs with a dosing regimen of approximately 2 weeks between infusion 1 and infusion 2, and 4 weeks between the remaining infusions.

SUMMARY:
This expanded access protocol is part of IND 027396 to evaluate efficacy and safety of multiple intravenous administrations of autologous HB-adMSCs for the treatment of Parkinson's disease for up to 11 patients who passed pre-screening, completed screening, and were not randomized into the treatment group for the HBPD03 clinical study protocol entitled, "A Randomized, Double-Blind, Single Center, Phase 2, Efficacy and Safety Study of autologous HB-adMSCs vs Placebo for the Treatment of Patients with Parkinson's Disease" under IND 027396.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have passed pre-screening for the HBPD03 clinical trial entitled, "A Randomized, Double-Blind, Single Center, Phase 2, Efficacy and Safety Study of autologous HB-adMSCs vs Placebo for the Treatment of Patients with Parkinson's Disease" under IND 027396.
2. Patients must have screened for the HBPD03 clinical trial entitled, "A Randomized, Double-Blind, Single Center, Phase 2, Efficacy and Safety Study of autologous HB-adMSCs vs Placebo for the Treatment of Patients with Parkinson's Disease" under IND 027396.
3. Patients must have not been randomized into the treatment group for the HBPD03 clinical trial entitled, "A Randomized, Double-Blind, Single Center, Phase 2, Efficacy and Safety Study of autologous HB-adMSCs vs Placebo for the Treatment of Patients with Parkinson's Disease" under IND 027396.
4. Male and female participants 18 - 80 years of age.
5. Patients must have been diagnosed with early and/or moderate Parkinson's disease at least 6 months before participation.
6. Patients must have previously banked their mesenchymal stem cells with Hope Biosciences.
7. Patients should be able to read, understand and to provide written consent.
8. Voluntarily signed informed consent obtained before any expanded access-related procedures are performed.
9. Female patients should not be pregnant or plan to become pregnant during participation and for 6 months after last investigational product administration.
10. Male patients if their sexual partners can become pregnant should use a method of contraception during participation and for 6 months after the last administration of the investigated product.
11. Patient is able and willing to comply with the requirements of this Expanded Access.

Exclusion Criteria:

1. Patients with advanced Parkinson's disease. Advanced PD is defined as a significant disability, wheelchair-bound or bedridden.
2. Any malignancy or clinical evidence that supports the presence of a malignant process in a patient is being investigated. Malignancy is defined as any form of cancer that had occurred in the previous five years before the first infusion and may require surgery, chemotherapy, or radiation.
3. Patients with medical history of uncontrolled high blood pressure defined as a deficient standard of care treatment and/or blood pressure > 150/90 mm/Hg during screening visit.
4. Patients with the following concomitant or past medical history:

   * Heart Failure - New York Heart Association (NYHA) Class III/IV.
   * Heart Attack (in the past six months before 1st infusion).
   * Stroke (in the past six months before 1st infusion).
   * Hepatitis B or C.
   * Human immunodeficiency virus (HIV) infection.
5. Any of the following abnormal lab findings during screening will disqualify a patient from this expanded access protocol:

   * Hemoglobin (Hgb) <10 G/DL or >18 G/DL
   * Hematocrit (HCT) <30% or >55%
   * Platelet count < 80 K/UL and or > 450 K/UL.
   * White blood cell count WBC < 3.0 K/UL and > 13.0 K/UL.
   * Alanine aminotransferase (ALT) of > 75 IU/L
   * Aspartate aminotransferase (AST) of > 75 IU/L
   * eGFR < 40 mL/min/1.73
   * Pre-prandial glucose > 150 MG/DL
   * Post-prandial glucose > 200 MG/DL
6. Patients who have received any stem cell treatment in the past six months before 1st infusion other than stem cells produced by Hope Biosciences.
7. Patients who are unlikely to complete the visits or adhere to the procedures.
8. The patient has previously been diagnosed with a psychiatric disorder, which is currently uncontrolled.
9. Patients with a history of addiction or dependency or currently abusing or using substances.
10. Patients with any form of kidney dialysis will be excluded from participation in the investigation.
11. Patients who have received an experimental drug in the past 12 months before the first dose of the investigational product. (Except for COVID-19 vaccinations).
12. Patients who the Investigator determines to be unsuitable for participation for other reasons, such as, but not limited to deep vein thrombosis (DVT), pulmonary embolus, cardiac arrhythmia, or those who have a prothrombotic condition, or who require persistent oxygen supplementation.
13. Patients who have recently undergone major surgery (in the past six months before 1st infusion). Some examples of major surgeries include, but are not limited to, the following: heart surgeries, aortic aneurysm bypass, organ transplant, intracranial surgery, spinal laminectomy or fusion, amputation, resection of the lung, resection of esophagus, resection of a mediastinal mass, resection of bladder or prostate tumor and resection of kidney or ureter.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Hope Biosciences Research Foundation